CLINICAL TRIAL: NCT01745978
Title: The Efficacy and Safety of Precut Papillotomy Using the Knob-tipped Knife and Needle Knife in Difficult Biliary Cannulation: a Randomized-controlled Trial.
Brief Title: Compare the Knob-tipped Knife With the Needle Knife in Difficult Biliary Cannulation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: changhai-121202
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography; Bile Duct Diseases
MeSH Terms: conditions — Bile Duct Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the knob-tipped knife (Experimental): the knob-tipped knife using for precut papillotomy in difficult CBD cannulation
  Interventions: Procedure: Precut papillotomy
- the needle knife (Active Comparator): the needle knife using for precut papillotomy in difficult CBD cannulation
  Interventions: Procedure: Precut papillotomy

INTERVENTIONS:
Procedure: Precut papillotomy

SUMMARY:
The aim of the present study was to compare the efficacy and safety of the knob-tipped knife and needle knife for precut papillotomy in difficult common bile duct (CBD)cannulation.

DETAILED DESCRIPTION:
Precut sphincterotomy is an alternative technique used to facilitate CBD cannulation following the failure of conventional bile duct cannulation. Needle knife papillotomy is the most widely practiced precut technique. However,Pre-cutting the papilla with a needle-knife is difficult, requiring experience and dexterity to control the axis and depth of the cut. Due to the increased rate of complications associated with this procedure, including pancreatitis, hemorrhage, and perforation, it was recommended to be performed only by experienced endoscopists.

The knob-tipped knife, a novel instrument utilizing a 2mm or 1.5mm cutting knife, is usually used for endoscopic submucosal dissection (ESD). Its knob-shaped tip and nonadjustable length make the knife less likely to slip and penetrate the tissue during the resection. Since the process of precut papillotomy is similar to ESD, the precutting procedure with the knob-tipped knife may be easier to be performed, as well as be safer. The efficacy and safety of this instrument in precut papillotomy have not been reported. We therefore assessed the efficacy and safety of the knob-tipped knife in precut papillotomy in difficult CBD cannulation.

ELIGIBILITY:
Inclusion Criteria:

* intact papilla and deep cannulation of the bile duct
* a standard wire-guided cannulation >10 minutes, OR Pancreatic contrast injections ≥3, OR Pancreatic deep wire pass ≥5

Exclusion Criteria:

* ampullary tumors
* Billroth II or Roux-en-Y anatomy
* prior endoscopic sphincterotomy(EST) or biliary stent
* choledochoduodenal fistulae

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Successful biliary cannulation rate after precut papillotomy | During endoscopic retrograde cholangiopancreatography (ERCP) procedure

SECONDARY OUTCOMES:
Biliary cannulation time after precut papillotomy | From precut papillotomy started to biliary cannulation achieved or abandoned

OTHER OUTCOMES:
The incidence of Early complications of endoscopic retrograde cholangiopancreatography(ERCP) including pancreatitis, hemorrhage, and perforation | 7 days after ERCP

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China